CLINICAL TRIAL: NCT02487004
Title: The Study of Association Between Intradialysis Sodium Balance and Clinical Outcomes in Chronic Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Su-Hyun Kim (Other)
Collaborators: Gambro Korea, LTD. (Industry)
Responsible Party: Sponsor-Investigator, Su-Hyun Kim, associate professor, Chung-Ang University
Organization: Chung-Ang University (Other)
Other Study IDs: CAU-1440
Record Dates: First submitted 2015-06-25; First posted 2015-07-01 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: End-stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Renal Dialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- chronic hemodialysis patients
  Interventions: Device: hemodialysis

INTERVENTIONS:
Device: hemodialysis

SUMMARY:
The purpose of this study is to determine whether the change of serum and dialysate sodium level during hemodialysis can influence on blood pressure and intradialytic weight gain in chronic hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* age 20 years or more
* hemodialysis vintage over 3 months
* dialyzed for 4 hours three times per week
* hemodialysis adequacy (Kt/V) over 1.2

Exclusion Criteria:

* diagnosed with chronic hepatitis or infection

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with end-stage renal disease requiring chronic hemodialysis
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
intradialytic sodium gradient | baseline and 4 hours
  change of serum sodium level between initiation and termination of hemodialysis

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ang University Hospital, Seoul, South Korea